CLINICAL TRIAL: NCT00522327
Title: Remote Simultaneous Medical Interpretation: Medical Outcomes
Brief Title: Remote Simultaneous Medical Interpreting and Medical Outcomes
Acronym: RSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: The California Endowment (Other); The Commonwealth Fund (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: Calendow/CMWF
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: DIabetes
Keywords: Immigrant; Interpreting
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): remote simult med interpret
  Interventions: Other: remote simultaneous medical interpreting
- 2 (Active Comparator): Usual & Customary
  Interventions: Other: usual and customary
- 3 (Other): comparison group
  Interventions: Other: ENglish speaking

INTERVENTIONS:
Other: remote simultaneous medical interpreting — remote simultaneous medical interpretation
  Arms: 1
Other: usual and customary — usual and customary interpreting
  Arms: 2
Other: ENglish speaking — English speakers
  Arms: 3

SUMMARY:
All new patients to the general medicine clinic who were not primarily English speaking were randomized, after consenting, to receieve either remote simultaneous medical interpreting or usual and customary interpreting services. Patient charts were followed for one year after enrollment to assess medical outcomes, including patient satisfaction, diabetes management, lipid management, depression screening and management, vaccine administration.

All Spanish-speaking ER patients were similarly enrolled. They were followed for one ER visit and their knowledge of exit instructions was assessed, as well as their satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* Limited English-speaking
* English-speaking
* New patient in medicine clinic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2004-11; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Adherence with care | one year

SECONDARY OUTCOMES:
care parameters | one year

CONTACTS AND LOCATIONS:
Overall Officials: Francesca M Gany, MD., M.S., Principal Investigator — NYU Langone Health

REFERENCES:
- [Derived] Leng JC, Changrani J, Gany FM. Language discordance and testing for latent tuberculosis infection among recent Asian and Latino immigrants. J Community Health. 2011 Apr;36(2):228-30. doi: 10.1007/s10900-010-9301-2. PMID 20697787
- [Derived] Leng JC, Changrani J, Tseng CH, Gany F. Detection of depression with different interpreting methods among Chinese and Latino primary care patients: a randomized controlled trial. J Immigr Minor Health. 2010 Apr;12(2):234-41. doi: 10.1007/s10903-009-9254-7. PMID 19408119
- [Derived] Gany F, Leng J, Shapiro E, Abramson D, Motola I, Shield DC, Changrani J. Patient satisfaction with different interpreting methods: a randomized controlled trial. J Gen Intern Med. 2007 Nov;22 Suppl 2(Suppl 2):312-8. doi: 10.1007/s11606-007-0360-8. PMID 17957417